CLINICAL TRIAL: NCT02897817
Title: Treatment Adherence in Patients With Rheumatoid Arthritis Previously Treated With Oral or Injectable Methotrexate and Requiring a New Treatment With Injectable Methotrexate
Brief Title: Treatment Adherence to Injectable Methotrexate in Rheumatoid Arthritis
Acronym: APRim
Status: Completed | Type: Observational
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: APRim
Record Dates: First submitted 2016-08-04; First posted 2016-09-13 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate; Treatment adherence
MeSH Terms: conditions — Arthritis, Rheumatoid; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oral to Injectable: Patients treated with oral MTX and requiring a switch to injectable MTX
- Injectable to Injectable: Patients treated with injectable MTX and eligible for a change in MTX injection device.

SUMMARY:
The aim of this study is to evaluate, at 6 months, the rate of patients whose adherence to injectable MTX remained strong or improved according to patient-reported outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Patients with a diagnosis of RA as confirmed by the ACR/EULAR (2010) Classification Criteria for Rheumatoid Arthritis
* Patients:

  * currently treated with oral MTX and requiring a switch to an injectable MTX* or
  * currently treated with an injectable MTX* and eligible for a change of MTX injection device*
* Patients informed about and accepting the computer processing of their medical data and their right of accesss and correction.

Exclusion Criteria:

- Patients who refuse to participate in the study or are unable to fill out the patient diary.

*On the basis of the products marketed at the time of submission of the study to Oversight Authorities (Méthotrexate Biodim®, Metoject® and imeth®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients currently treated with oral methotrexate (MTX) and requiring a switch to injectable MTX or currently treated with an injectable MTX and eligible for a change to a different MTX injection device will be asked to participate from RA treatment change (inclusion visit) up to 6 months after inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rate of patients whose adherence to methotrexate (MTX) remained strong or improved between inclusion (V0) and follow-up (V1) at 6 months. | 6 months
  Patient adherence is measured via the Morisky score at V0 and V1, using patient-reported outcome (PRO).

SECONDARY OUTCOMES:
Comparison of patient adherence between the 2 cohorts. | 6 months after inclusion.
  Analysis of improved or equivalent patient adherence as assessed by the Morisky score at V0 and V1 between the 2 cohorts.
Reasons for non-adherence given by patients after 6 months. | 6 months after inclusion.
  Assessed in the overall patient population and between the 2 cohorts.
Global and functional patient satisfaction with treatment after 6 months as assessed by the Likert scale for global satisfaction. | 6 months after inclusion.
  Global patient satisfaction will be assessed in the overall patient population and between the 2 cohorts using the Likert scale (1 to 5 rating).
Global and functional patient satisfaction with treatment after 6 months as assessed by the Disease Activity Score 28 (DAS28) for disease severity. | 6 months after inclusion.
  Patient satisfaction will be assessed in the overall patient population and between the 2 cohorts using the DAS28.
Global and functional patient satisfaction with treatment after 6 months as assessed by the Health Assessment Questionnaire Disability Index (HAQ-DI) for functional disability. | 6 months after inclusion.
  Patient satisfaction will be assessed in the overall patient population and between the 2 cohorts using the HAQ-DI.
Global and functional patient satisfaction with treatment after 6 months as assessed by the Echelle de Mesure de l'Impact de la polyarthrite Rhumatoïde (EMIR) for quality of life. | 6 months after inclusion.
  Patient satisfaction will be assessed in the overall patient population and between the 2 cohorts using the EMIR.
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on family situation. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing family situation. Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on socio-professional standing. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing socio-professional standing. Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on age. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing age. Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on comorbidities. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing comorbidities. Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on the co-administration of other injectable treatments. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing the co-administration of other injectable treatments (binary variable). Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on the reasons for the switch to new MTX injection device. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing the reasons for the switch to new MTX injection device. Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the change in the Morisky scores at V0 and V1, based on rheumatoid arthritis severity (assessed by DAS28). | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing rheumatoid arthritis severity (assessed by DAS28). Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, evaluated by the change in the Morisky scores at V0 and V1, based on patient functional handicap (assessed by the HAQ-DI). | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing functional handicap (assessed by the HAQ-DI). Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, as evaluated by the Morisky score at V0 and V1, based on global patient satisfaction (assessed by Likert scale results). | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing global patient satisfaction (assessed by Likert scale results). Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, evaluated by the change in the Morisky scores at V0 and V1, based on whether the injection was self-administered or administered by a third party. | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing whether the injection was self-administered or administered by a third party. Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Analysis of improvement or maintenance of patient adherence, evaluated by the change in the Morisky scores at V0 and V1, based on tolerability and level of patient trust with HCP (assessed by Likert scale results). | 6 months after inclusion.
  Identification of factors associated with the improvement or maintenance of adherence in the overall patient population and between the 2 cohorts by assessing tolerability and level of patient trust with HCP (assessed by Likert scale results). Adherence is evaluated by the change in the Morisky scores at V0 and V1, with a score of 0 considered as strong adherence and a score >0 considered as non-adherence. Patient adhesion is classified as remaining strong if the Morisky score at V0 and V1 remains at 0 and patient adhesion is classified as improved if the Morisky score at V0 is greater than 0 (non-adherent) while the score at V1 is 0 (strong adherence).
Doctor satisfaction with the treatment after 6 months. | 6 months after inclusion.
  Assessed in the overall patient population and between the 2 cohorts.
Treatment adherence, evaluated by the Morisky score at 6 months, as assessed by the HCP compared to the treatment adherence as reported by the patient . | 6 months after inclusion.
  Treatment adherence is measured via the Morisky score at V0 and V1.

CONTACTS AND LOCATIONS:
Overall Officials: René-Marc FLIPO, MD, Prof, Principal Investigator — CHU Hôpital Roger Salengro, LILLE; Eric SENBEL, MD, Principal Investigator — Doctor's Office, MARSEILLE; Sonia TROPE, Nurse, Principal Investigator — ANDAR; Hélène HERMAN-DEMARS, MD, Study Director — NORDIC PHARMA
Locations (1):
- Nordic Pharma, Paris, France